CLINICAL TRIAL: NCT03488264
Title: Understanding the Intersection of Stigma and Self-Management of Sickle Cell Disease
Brief Title: Stigma, Self-management, & Quality of Life in SCD
Acronym: SSQ
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00084001
Record Dates: First submitted 2018-03-29; First posted 2018-04-04 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-03

CONDITIONS: Sickle Cell Disease; Quality of Life; Stigma, Social; Disease Self-Management
MeSH Terms: conditions — Anemia, Sickle Cell; Social Stigma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- United States: 50 participants will be recruited from the United States.
- Jamaica: 50 participants will be recruited from Jamaica.

SUMMARY:
Many individuals with sickle cell disease experience both a poor quality of life and stigma. Individuals with SCD often experience high levels of stigma which can be a barrier to good self-management and hinder quality of life. The purpose of this research is to improve understanding of the relationships between stigma, self-management, and quality of life in SCD in the United States and Jamaica. The findings from this project will contribute to the development of a tool to measure self-management strategies and will also guide the development of interventions to improve SCD self-management.

DETAILED DESCRIPTION:
The goal of the proposed study is to explore the complex relationships between perceived stigma, demographic and clinical characteristics, sickle cell disease (SCD) self-management strategies, and quality of life (QoL) in adults with SCD in the United States (US) and Jamaica, countries with important differences relevant to this study. Proposed is a cross sectional study that will use a convergent parallel mixed methods design (individual interviews and self-report surveys). Participants will be interviewed about SCD self-management strategies and how sources of stigma influence these strategies. Quantitative measures will be used to assess perceived stigma [SCD Health-Related Stigma Scale (SCD-HRSS)] and QoL [Adult Sickle Cell Quality of Life Measures (ASCQ-Me): emotional impact, pain episodes, pain impact, sleep impact, social functioning impact, and stiffness impact; disease severity]. The primary outcome of the study is stigma and the secondary outcome is QoL(emotional impact, pain episodes, pain impact, sleep impact, social functioning impact, and stiffness impact; disease severity).

The specific aims of this study are to:

Aim 1: Determine the influences of perceived stigma and demographic and clinical characteristics on SCD self-management and QoL in adults with SCD in the US and Jamaica.

Question 1: What are the influences of perceived stigma and demographic and clinical characteristics on SCD self-management? Question 2: What are the influences of perceived stigma and demographic and clinical characteristics on QoL? Aim 2: Describe the relationship between SCD self-management strategies and QoL.

ELIGIBILITY:
Inclusion Criteria:

1. at least 18 years of age,
2. ability to understand English,
3. diagnosis of SCD based on one of the following genotypes (ICD-10-CM code): HbSS (D57.0-D57.02), HbSC (D57.2-57.21), Hb SS/Bthalassemia+ or Hb SS/a-thalassemia- (D57.1, D57.4-D57.41, D57.8-D57.819).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with sickle cell disease in the United States and Jamaica
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2018-10-27 (Actual); Study Completion 2018-10-27 (Actual)

PRIMARY OUTCOMES:
Health-Related Stigma | 10 minutes
  The Sickle Cell Disease Health-Related Stigma Scale (SCD-HRSS) will assess stigma. SCD-HRSS has 4 subscales that measure stigma from the public, doctors, nurses, and family; and consists of 40 items on a 6 point Likert scale. It is scored by obtaining the sum of the mean score of the four subscales (subscales: 10-60; total scale: 40-240). Higher scores indicate higher perceived stigma.
Disease-related Stigma | 5 minutes
  The Measure of Sickle Cell Stigma (MoSCS) will assess stigma. MoSCS consists of 11-items with 4 subscales assessing social exclusion, internalized stigma, disclosure concerns, and expected discrimination. It is measured on a 6 point Likert scale; scores range from 6-36 and are obtained by summing and averaging the total scale. Higher scores indicate higher perceived stigma.

SECONDARY OUTCOMES:
Quality of life | 14-21 minutes
  Quality of life will be measured using Adult Sickle Cell Quality of life Measures (ASCQ-Me) subscales for emotional impact, pain episodes, pain impact, sleep impact, social functioning impact, and stiffness impact. For pain episodes separate composite scores are calculated for pain frequency (0-11) and severity (0-22). Higher scores indicate worse health status. Raw scores for the remaining scales range 5-25 and are developed by using T-Score transformation to standardize raw scores to have a mean of 50 (indicates an average health score on the scale) and standard deviation of 10 (represents one SD). Higher scores indicate healthier status.
Emotional impact | 2-3 minutes
  Score on the ASCQ-Me Emotional Impact - Raw scores for this scale ranges 5-25 and are developed by using T-Score transformation to standardize raw scores to have a mean of 50 (indicates an average health score on the scale) and standard deviation of 10 (represents one SD). Higher scores indicate healthier status.
Pain episodes | 2-3 minutes
  Score on ASCQ-Me Pain episodes - For pain episodes separate composite scores are calculated for pain frequency (0-11) and severity (0-22). Higher scores indicate worse health status.
Pain impact | 2-3 minutes
  Score on ASCQ-Me Pain impact - Raw scores for this scale ranges 5-25 and are developed by using T-Score transformation to standardize raw scores to have a mean of 50 (indicates an average health score on the scale) and standard deviation of 10 (represents one SD). Higher scores indicate healthier status.
Sleep impact | 2-3 minutes
  Score on ASCQ-Me Sleep impact - Raw scores for this scale ranges 5-25 and are developed by using T-Score transformation to standardize raw scores to have a mean of 50 (indicates an average health score on the scale) and standard deviation of 10 (represents one SD). Higher scores indicate healthier status.
Social functioning impact | 2-3 minutes
  Score on ASCQ-Me Social functioning impact - Raw scores for this scale ranges 5-25 and are developed by using T-Score transformation to standardize raw scores to have a mean of 50 (indicates an average health score on the scale) and standard deviation of 10 (represents one SD). Higher scores indicate healthier status.
Stiffness impact | 2-3 minutes
  Score on the ASCQ-Me stiffness impact - Raw scores for this scale ranges 5-25 and are developed by using T-Score transformation to standardize raw scores to have a mean of 50 (indicates an average health score on the scale) and standard deviation of 10 (represents one SD). Higher scores indicate healthier status.
Disease Severity | 2-3 minutes
  The ASCQ-Me Medical History Checklist (SCD-MHC) contains 9 items that list treatments and conditions associated with SCD (leg ulcers, avascular necrosis) that are scored dichotomously (0-9) with higher scores indicating higher disease severity.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Tanabe, PhD, Principal Investigator — Duke University
Locations (2):
- Dominique Bulgin, Durham, North Carolina, United States
- Sickle Cell Unit, The University of the West Indies, Mona, Kingston 7, Jamaica

IPD SHARING:
Plan to Share IPD: No